CLINICAL TRIAL: NCT02657135
Title: Targeted Evaluation, Action, & Monitoring of Traumatic Brain Injury
Acronym: TEAM-TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Okonkwo, MD, Phd, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: W81XWH-14-2-0002
Record Dates: First submitted 2015-07-16; First posted 2016-01-15 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Traumatic Brain Injury (TBI)
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Neuropsychological Tests; Magnetic Resonance Spectroscopy; Magnetoencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- History of Traumatic Brain Injury (Experimental): All participants have a history of TBI. At study outcome participants are provided treatment recommendations that are the result of a consensus meeting of all physician investigators. Follow up care is not provided by this clinical trial.
  Interventions: Behavioral: Cognitive/Neuropsychological Testing; Other: Vestibular/Ocular-Motor Testing; Other: Cervical (Neck) Evaluation; Other: Sleep Evaluation; Other: HDFT MRI; Other: MR Spectroscopy (MRS); Other: MEG (Magnetoencephalography)

INTERVENTIONS:
Behavioral: Cognitive/Neuropsychological Testing — These tests will be used to determine how the participant will continue with future procedures, and depending on results, may involve the participant returning to complete subsequent testing.
Other: Vestibular/Ocular-Motor Testing — These assessments will involve a series of tests and questionnaires that focus on physical symptoms of TBI and will include dizziness, balance, ocular-motor coordination, and reflexes.
Other: Cervical (Neck) Evaluation — These assessments will involve a series of tests and questionnaires that focus on physical symptoms of TBI including neck mobility and pain levels.
Other: Sleep Evaluation — These evaluations will focus on assessing insomnia (duration, frequency, daytime consequences), combat exposure, and the presence and severity of trauma history.
Other: HDFT MRI — This MRI aims at providing qualitative and quantitative assessments of the nature, location, and extent of white matter injury.
Other: MR Spectroscopy (MRS) — This is a noninvasive diagnostic test for measuring biochemical changes in the brain.
Other: MEG (Magnetoencephalography) — This is a non-invasive neurophysiological technique that measures the magnetic fields generated by neuronal activity of the brain.

SUMMARY:
TEAM-TBI (Targeted Evaluation, Action, and Monitoring of Traumatic Brain Injury) is a research study that brings together TBI patients, advanced evaluation methods, and experts in a multi-faceted study to address the heterogeneity of TBI and to evaluate the effects self-help strategies might have on TBI outcomes.

DETAILED DESCRIPTION:
TEAM-TBI (Targeted Evaluation, Action, and Monitoring of Traumatic Brain Injury) proposes a new approach to clinical trials in TBI that will:

* Evolve diagnostic technology & treatment
* Improve self-help strategies
* Lower cost and speed for delivery of effective strategies

The TEAM-TBI program proposes an innovative new approach to TBI clinical trials to overcome the limitations of past efforts and achieve long-awaited breakthroughs for TBI survivors. The study will involve a comprehensive 3-4 day intake evaluation, followed by a variety of remotely performed tasks during a 1-6 month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age
* Fluent in English
* Documented history of TBI or blast exposure since 2001

Exclusion Criteria:

* Inability to have MRI
* Pregnancy
* History of TIA within last 6 months.
* Presently involved in open litigation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2014-03-24 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
The main outcome variable in the study will be the change in Post-Concussion Symptom Scale (PCSS) score from the initial intake evaluation compared to last follow-up evaluation. | Up to 6 months

SECONDARY OUTCOMES:
Change in the Satisfaction with Life Scale | Up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Neurotrauma Clinical Trials Center, Pittsburgh, Pennsylvania, United States